CLINICAL TRIAL: NCT05530694
Title: Implementation of Shared Decision Making in Rheumatoid Arthritis: A Stepped Wedge, Cluster-randomized Trial
Brief Title: Rheumatoid Arthritis Shared Decision Making
Acronym: RAiSeD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 20-162
Record Dates: First submitted 2022-07-21; First posted 2022-09-07 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Rheumatoid Arthritis
Keywords: shared decision making; rheumatoid arthritis; rheumatology
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: Stepped wedge cluster randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Usual care
- Intervention (Experimental): Intervention phase
  Interventions: Behavioral: Clinician communication training; Behavioral: Patient activation; Behavioral: RA Medication summary guide and RA Choice

INTERVENTIONS:
Behavioral: Clinician communication training — The clinician training is a generic, skills- and attitude-based approach for clinicians to acknowledge their decision making conversations with patients that 1) there is more than one option, and 2) patient's views matter in deciding what to do next. This tools-free approach can be used on the spot when needed and is termed fostering choice awareness (FCA). The one-hour training consists of 4 parts: 1) a knowledge session on evidence and guidelines on effective conversations and SDM, 2) video-review of behaviors which foster or hinder choice awareness, 3) clinical simulations in which clinicians practice fostering choice awareness behaviors, and 4) a reminder card for use in future clinic visits. Video clips will be of patient-clinician conversations around treatment decision making to prompt and probe clinicians' experiences, improve understanding, and improve practice.
  Other Names: fostering choice awareness
  Arms: Intervention
Behavioral: Patient activation — The patient activation component consists of three questions patients can ask their clinician to help them become more involved: "1. What are my options?; 2. What are the possible benefits and harms of those options?; 3. How likely are each of those benefits and harms to happen to me?" These questions have been used in studies to promote improved communication in a number of conditions including cardiovascular disease, cancer, and women's health.
  Other Names: AskShareKnow
  Arms: Intervention
Behavioral: RA Medication summary guide and RA Choice — RA Choice presents information on FDA-approved RA treatments in a set of cards, which can be used alone or in combination based on a patient's preference, values, and the clinician's experience. The RA medication summary guide describes options for medication, physical therapy, occupational therapy, and ways to stay healthy with diet and exercise. Tool development followed key principles of creating low literacy materials that featured icons, short phrases written in plain language, and included topics of interest to RA patients faced with a medication decision. For the proposed study, we will include a paper-based version of the tool, or a web-based version available for telephone or VA Video Connect (VVC) visits. The tools will be updated to include new FDA-approved therapies (e.g., JAK inhibitors).
  Arms: Intervention

SUMMARY:
Shared decision making is the first overarching principle for the treat to target guidelines for rheumatoid arthritis (RA) and has been proposed as a potential mechanism to reduce health disparities, however there is little evidence to inform effective ways to implement this practice in the care of Veterans with RA. The purpose of this project is to evaluate the effectiveness of a multi-component shared decision making intervention on RA disease activity, adherence to RA medications and patient knowledge of RA. The proposed research will contribute to fundamental knowledge about how to effectively foster shared decision making across varied VA rheumatology clinical settings to improve patient disease outcomes and experience; and support clinicians to engage patients in meaningful ways with the ultimate goal to improve health, reduce disability, and eliminate disparities.

DETAILED DESCRIPTION:
Background: Rheumatoid arthritis (RA) impacts quality of life causing disability in up to 1% of the population and 2% of those 60 and older. Men with RA have twice the risk of death as the general population. Treatment decisions after failure with first-line methotrexate are complex, involve trade-offs in terms of harm, and require individualized decisions. In shared decision making (SDM), patients and clinicians work together to identify how to best address the patient's situation. SDM has been proposed as a way to reduce disparities, but uptake is suboptimal and no effective tools to foster SDM in a systematic way across VA exist.

Significance/Impact: Veterans with RA are disproportionately male, have more comorbidities, and higher mortality rates in comparison to the general population. SDM is the first principal of the RA treat to target guidelines. However, significant gaps in knowledge of effective interventions to support SDM exist - particularly in VA. This proposal is responsive to three VA HSR&D priority domains: 1) health care value, 2) quality of health care, and 3) health equity.

Innovation: Treatment studies in RA have focused primarily on white women, while men, who represent the VA RA population, have poorer outcomes. Targeting this subgroup to evaluate the impact of an SDM intervention on disease outcomes and adherence is novel. Use of a novel approach combining clinician training and a decision aid to recognize the unique needs of Veterans with RA is innovative.

Specific Aims: Aim 1: Evaluate the effectiveness of a multi-component SDM intervention in a stepped-wedge, cluster-randomized controlled trial on improvement in disease activity, RA knowledge, and adherence. Hypothesis 1: During SDM intervention phases, Veterans will have lower disease activity compared to during control periods and will be more likely to experience clinically important differences in a standard disease activity index. Hypothesis 2: Veterans will have greater RA knowledge and better adherence after exposure to this intervention. Exploratory Hypothesis: The SDM intervention will have a greater effect in the likelihood of lowering disease activity among racial/ethnic minorities and Veterans with limited health literacy. Aim 2: Evaluate effectiveness of a multi-component intervention to facilitate SDM. Hypothesis: An SDM intervention for Veterans with RA will result in higher uptake of SDM in enrolled clinics during the intervention phase, relative to control phase. Aim 3: Conduct a qualitative evaluation of the SDM intervention and local implementation to inform future dissemination.

Methodology: A stepped-wedge, cluster-randomized controlled trial design will be used to evaluate effectiveness of a novel SDM intervention across three sites. Participants: Veterans with RA and rheumatology clinicians; Intervention: multicomponent SDM intervention ; Control: participants at each site during the pre-intervention period; Outcomes: RA disease activity; patient-reported measures of adherence, knowledge, SDM, and an objective measure of SDM. Time: pre-intervention, intervention, and post-intervention phases for each step, measures collected over 42 months.

Implementation/Next Steps: The proposed effectiveness study has the potential to speed the translation of SDM research within VA and nationally to improve quality of care for all persons with RA.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for patient participants (Aims 1 & 2):

* Meet administrative data definition of rheumatoid arthritis (see recruitment section)
* Receive rheumatology outpatient care at participating clinics and seen at least once in prior 12 months
* Age 18 years or older
* English speaking
* Moderate to high RA disease activity within 18 months prior to enrollment

Inclusion criteria for professional participants (Aims 1-3):

-Rheumatology attendings, fellows or advanced practice partners (nurse practitioners or physicians assistants) at the respective clinics

Inclusion criteria for non-clinician participants (Aim 3):

* Have held a leadership position within their respective institution for minimum of 12 months prior to enrollment
* Have worked in the rheumatology clinic setting at their respective institution for minimum of 12 months prior

Exclusion Criteria:

Exclusion criteria for patient participants (Aims 1 & 2):

* Cognitive impairment
* Inability to speak

Exclusion criteria for professional participants (Aims 1-3):

-none

Exclusion criteria for non-clinician participants (Aim 3):

* Have held a leadership position within their respective institution for <12 months
* Have worked in a clinic setting other than rheumatology
* Have worked in a clinic setting <12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 792 (Estimated)
Dates: Start 2022-09-19 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Disease activity | through study completion (up to 4 years), on average 3 times per year
  RA disease activity will be measured using composite score: the Clinical Disease Activity Index (range 0-76) or CDAI. This is a composite score of clinician assessed swollen and tender joints counts, clinician global assessment and patient global assessment of disease activity. Higher score is indicative of higher disease activity.

SECONDARY OUTCOMES:
Change in rheumatoid arthritis knowledge | measured at baseline, 6 months and 12 months on a subset
  Patient general knowledge of RA and RA medications will be measured using a 8-item self-reported survey. This measure is designed to capture rudimentary knowledge of RA and RA medications. A score of 7 out of 8 correct answers is considered adequate RA knowledge. One or more missed dose per week is considered poor adherence.
Change in adherence | measured at baseline, 6 months and 12 months on a subset
  Patient-reported RA medication adherence will be assessed using a validated single-item measure: "How many times do you think you may have missed taking your pills in the last week?". A response of 1 or greater is considered nonadherent. Among participants taking a biologic therapy (self-injection or infusion), adherence will be measured asking, "How many times do you think you have missed your RA injection or infusion in the past month?" Adherence will be dichotomized into either poor or adequate adherence, with poor adherence defined as missing 1 RA pills over the past week or 1 RA injections in the past month.
CollaboRATE questionnaire | through study completion (up to 4 years), on average 3 times per year
  CollaboRATE is a brief, validated patient-reported 3-item measure to assess the process of shared decision making. Each item represents a dimension of shared decision making (explanation or the health issue, elicitation of patient preferences, and Integration of patient preferences). The questions are each rated on a 10-point anchored scale from 1 (no effort was made) to 10 (every effort was made). Higher scores indicate a better shared decision making experience.
Change in OPTION-5 (objective measure of shared decision making) | through study completion (up to 4 years), on average 1 time per year
  OPTION-5 is a measure of direct observation (audio-taped recordings) of shared decision making. The measure contains 5 items scored from 0 (absence of shared decision making) to 4 (optimal performance). A trained external observer will score the clinician on the extent to which they involve the patient in decision making, scores are summed and scaled to fall between 0-100 for ease of interpretation. Higher scores indicate greater uptake of shared decision making.
SURE questionnaire | through study completion (up to 4 years), on average 3 times per year
  SURE is a brief, validated patient-reported 4-item measure to assess patient uncertainty about treatment choice including uncertainty about benefits and risks, what matters most to the patient, support in making the choice, and feeling sure about the best choice. Patients rate each item true or false and scores can range from 0-4. A score below 4 is indicates decisional conflict and a score of 3 or less is considered clinically relevant decisional conflict.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Barton, MD, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (4):
- United States (4):
  - San Francisco VA Medical Center, San Francisco, CA, San Francisco, California
  - Wilmington VA Medical Center, Wilmington, DE, Wilmington, Delaware
  - VA Portland Health Care System, Portland, OR, Portland, Oregon
  - Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barton JL, Markwardt S, Niederhausen M, Schue A, Dougherty J, Katz P, Saha S, Yelin EH. Are We on the Same Page? A Cross-Sectional Study of Patient-Clinician Goal Concordance in Rheumatoid Arthritis. Arthritis Care Res (Hoboken). 2023 Mar;75(3):625-633. doi: 10.1002/acr.24794. Epub 2022 Nov 16. PMID 34569172
- [Background] Morrison T, Foster E, Dougherty J, Barton J. Shared decision making in rheumatology: A scoping review. Semin Arthritis Rheum. 2022 Oct;56:152041. doi: 10.1016/j.semarthrit.2022.152041. Epub 2022 Jun 3. PMID 35738040
- [Background] Hulen E, Larsen C, Matsumoto R, Katz P, Barton JL. "You can't touch, you can't bond": Exploring COVID-19 pandemic impacts on rheumatoid arthritis patient goals and communication with clinicians. Musculoskeletal Care. 2023 Mar;21(1):244-248. doi: 10.1002/msc.1689. Epub 2022 Sep 8. No abstract available. PMID 36073563
- [Background] Singh N, Grivas P, Makris UE, Suarez-Almazor ME, O'Hare AM, Barton JL. Use of Disease-Modifying Antirheumatic Drugs in Rheumatoid Arthritis: Supporting Shared Decision-Making Between Patients With Cancer and Clinicians. ACR Open Rheumatol. 2023 Jun;5(6):305-307. doi: 10.1002/acr2.11552. Epub 2023 May 11. No abstract available. PMID 37166652
- [Background] Baker R, Mantilla B, Graf J, Katz PP, Goglin S, Barton JL, Liew JW, Wysham KD. Racial and Ethnic Differences in a Biochemical Marker of Rheumatoid Arthritis Disease Activity. ACR Open Rheumatol. 2023 Mar;5(3):142-148. doi: 10.1002/acr2.11524. Epub 2023 Feb 8. PMID 36754575
- [Background] McGoldrick J, Molina-Ochoa D, Schwab P, Edwards ST, Barton JL. An Evaluation of Burnout Among US Rheumatology Fellows: A National Survey. J Rheumatol. 2023 Sep;50(9):1185-1190. doi: 10.3899/jrheum.221114. Epub 2023 Mar 15. PMID 36921966
- [Background] England BR, Smith BJ, Baker NA, Barton JL, Oatis CA, Guyatt G, Anandarajah A, Carandang K, Chan KK, Constien D, Davidson E, Dodge CV, Bemis-Dougherty A, Everett S, Fisher N, Fraenkel L, Goodman SM, Lewis J, Menzies V, Moreland LW, Navarro-Millan I, Patterson S, Phillips LR, Shah N, Singh N, White D, AlHeresh R, Barbour KE, Bye T, Guglielmo D, Haberman R, Johnson T, Kleiner A, Lane CY, Li LC, Master H, Pinto D, Poole JL, Steinbarger K, Sztubinski D, Thoma L, Tsaltskan V, Turgunbaev M, Wells C, Turner AS, Treadwell JR. 2022 American College of Rheumatology Guideline for Exercise, Rehabilitation, Diet, and Additional Integrative Interventions for Rheumatoid Arthritis. Arthritis Care Res (Hoboken). 2023 Aug;75(8):1603-1615. doi: 10.1002/acr.25117. Epub 2023 May 25. PMID 37227116
- [Background] Barton JL. Unequal Treatment: Physical Therapy Utilization in Rheumatoid Arthritis. J Rheumatol. 2023 Nov;50(11):1359-1361. doi: 10.3899/jrheum.2023-0814. Epub 2023 Sep 15. No abstract available. PMID 37714545
- [Background] Nasrallah C, Schmajuk G, Hamblin A, Wilson C, Kersey E, Young C, Katz P, Bajaj P, Downey C, Bartels C, Zell J, Danila MI, Ferguson S, Barton JL, DeQuattro K, Yazdany J. Leveraging the Consolidated Framework for Implementation Research to Develop the American College of Rheumatology's Toolkit for Implementation of Rheumatoid Arthritis Outcome Measures in Clinical Practice: A Qualitative Study. Arthritis Care Res (Hoboken). 2024 Dec;76(12):1647-1656. doi: 10.1002/acr.25410. Epub 2024 Sep 5. PMID 39099213
- [Background] Decary S, de Wit M, Naye F, Barton JL, Fraenkel L, Li LC, Brooks P, Stacey D, Maxwell LJ, Campbell W, Hofstetter C, Voshaar M, Meara A, Christensen R, Boonen A, Suarez-Almazor ME, Meade T, March L, Jull JE, Alten R, Morgan EM, Stewart Hazlewood G, Barber CEH, Guillemin F, El-Miedany Y, Mittoo S, Robertson TW, Bartlett SJ, Singh JA, Mannion M, Nasef SI, Boel A, Adebajo A, Arnaud L, Gill TK, Moholt E, Burt J, Jayatilleke A, Hmamouchi I, Berthelsen DB, Blanco FJ, Mather K, Maharaj A, Sharma S, Caso F, Beaton D, Shea B, Fong C, Fernandez AP, Mackie S, Nikiphorou E, Jones A, Greer-Smith R, Sloan VS, Akpabio A, Strand V, Lee RR, Umaefulam V, Monti S, Abaza N, Schultz G, Stones S, Gossec L, Nielsen SM, Cavallo S, Srinivasalu H, Constien D, Evans V, Tugwell P, Toupin-April K. Consensus on the definitions and descriptions of the domains of the OMERACT Core Outcome Set for shared decision making interventions in rheumatology trials. Semin Arthritis Rheum. 2024 Apr;65:152381. doi: 10.1016/j.semarthrit.2024.152381. Epub 2024 Jan 15. PMID 38306813
- [Background] Maxwell LJ, Wright GC, Schultz G, Grosskleg S, Barton JL, Campbell W, Guillemin F, Hofstetter C, Shea BJ, Simon LS, Adebajo A, Barnabe C, Goel N, Hurley P, Nikiphorou E, Petkovic J, Tugwell P. Embracing unity at OMERACT: Valuing equity, promoting diversity, fostering inclusivity. Semin Arthritis Rheum. 2024 Jun;66:152422. doi: 10.1016/j.semarthrit.2024.152422. Epub 2024 Feb 29. PMID 38461757
- [Background] Naye F, Toupin-April K, de Wit M, LeBlanc A, Dubois O, Boonen A, Barton JL, Fraenkel L, Li LC, Stacey D, March L, Barber CEH, Hazlewood GS, Guillemin F, Bartlett SJ, Berthelsen DB, Mather K, Arnaud L, Akpabio A, Adebajo A, Schultz G, Sloan VS, Gill TK, Sharma S, Scholte-Voshaar M, Caso F, Nikiphorou E, Nasef SI, Campbell W, Meara A, Christensen R, Suarez-Almazor ME, Jull JE, Alten R, Morgan EM, El-Miedany Y, Singh JA, Burt J, Jayatilleke A, Hmamouchi I, Blanco FJ, Fernandez AP, Mackie S, Jones A, Strand V, Monti S, Stones SR, Lee RR, Nielsen SM, Evans V, Srinivasalu H, Gerard T, Demers JL, Bouchard R, Stefan T, Dugas M, Bergeron F, Beaton D, Maxwell LJ, Tugwell P, Decary S. OMERACT Core outcome measurement set for shared decision making in rheumatic and musculoskeletal conditions: a scoping review to identify candidate instruments. Semin Arthritis Rheum. 2024 Apr;65:152344. doi: 10.1016/j.semarthrit.2023.152344. Epub 2023 Dec 16. PMID 38232625
- [Background] England BR, Smith BJ, Baker NA, Barton JL, Oatis CA, Turner AS. Reply. Arthritis Care Res (Hoboken). 2024 Mar;76(3):438-439. doi: 10.1002/acr.25255. Epub 2023 Dec 17. No abstract available. PMID 37818722
- [Background] Schue A, Matsumoto R, Barton J. Goal Concordance in Rheumatoid Arthritis Patients with Depression - What Do Patients Prioritize? [Abstract]. Arthritis & rheumatology (Hoboken, N.J.). 2023 Nov 14; 75(Suppl 9):2032.
- [Derived] Barton JL, Niederhausen M, Tuepker A, Schmajuk G, Baker J, Lovejoy TI, Morasco BJ, Kunneman M, Scholl I. Implementation of shared decision making in rheumatoid arthritis: study protocol for RAiSeD (Rheumatoid Arthritis Shared Decision Making) stepped wedge, cluster-randomized trial. Trials. 2025 Sep 29;26(1):381. doi: 10.1186/s13063-025-09015-1. PMID 41024266